CLINICAL TRIAL: NCT01122394
Title: Reducing Risk of Recurrences: Issues in Maintenance and Stability in Stroke (CDA 08-009)
Brief Title: Reducing Risk of Recurrence
Acronym: RRR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDP 09-414
Record Dates: First submitted 2010-05-10; First posted 2010-05-13 (Estimated); Results first posted 2016-10-20 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-08

CONDITIONS: Stroke; TIA; Hypertension; Hyperlipidemia
Keywords: stroke; recurrence; blood pressure; prevention
MeSH Terms: conditions — Stroke; Hypertension; Hyperlipidemias; Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored Intervention (TI) (Experimental): Tailored intervention based on the transtheoretical model
  Interventions: Behavioral: TI
- Attention Placebo (AP) (Placebo Comparator): Attention Placebo
  Interventions: Behavioral: AP

INTERVENTIONS:
Behavioral: TI — Tailored intervention based on the transtheoretical model
  Arms: Tailored Intervention (TI)
Behavioral: AP — Attention placebo
  Arms: Attention Placebo (AP)

SUMMARY:
Adults who have had a previous stroke or transient ischemic attack (TIA) remain at risk for having a second serious event, especially if they have uncontrolled blood pressure or cholesterol. However, many patients have difficulty following treatment recommendations for lowering blood pressure and cholesterol. The purpose of this research project is to evaluate the effect of 2 booster sessions of an educational counseling intervention on how well adults who have already participated in a 6-month clinical trial had a stroke or transient ischemic attack (TIA) are able to follow a treatment plan and control their blood pressure and cholesterol levels. We will also examine how effective this intervention is in improving adherence to diet, medication, and physical activity recommendations for adults who have had a prior stroke or TIA.

DETAILED DESCRIPTION:
National recommendations state that patients with a history of transient ischemic attack (TIA) or ischemic stroke should receive hypertension treatment, including antihypertensive medication and lifestyle modification, with a goal of reducing blood pressure (BP) to <120 mm Hg systolic BP and <80 mm Hg diastolic BP. Statin treatment and lifestyle modification is also recommended for post-stroke and post-TIA patients with elevated cholesterol levels or a history of stroke or TIA with an atherosclerotic cause. Despite the clear benefits of secondary stroke prevention, there is a gap between evidence and implementation in clinical practice. We will determine whether a telephone-delivered behaviorally tailored intervention (TI) can lead to sustained change resulting in (a) BP and lipid control and (b) improved adherence to diet, medication, and exercise recommendations in veterans with a history of stroke or TIA compared to an attention placebo (AP) in veterans who have completed 6 months of a clinical trial. In this CDA project, we evaluate the long-term effectiveness of booster sessions in a randomized manner. One arm will receive 6 months of a tailored intervention (TI) followed by two booster TI sessions at 8 and 10 months, and one arm will receive 6 months of an attention placebo (AP) followed by two booster AP sessions at 8 and 10 months. BP (3 measures taken at least 5 min apart) and dietary sodium are the primary outcomes, while secondary outcomes will be total cholesterol/high density lipoprotein ratio, adherence to antihypertensive and lipid-lowering drugs, and exercise adherence.

ELIGIBILITY:
Inclusion Criteria:

* Well-documented history of stroke or TIA that occurred at least 3 months prior to enrollment;
* Age 21 years or older;
* Continuity of care in the VAMC primary care or neurology clinics, defined as at least 1 visit in either clinic during the past 1 year;
* On hypertensive and/or lipid-lowering agents;
* A score of >16 on the Mini-Mental Status Exam;
* ability to exercise (assessed by 6-minute walk or timed get up and go).

Exclusion Criteria:

* Limited life expectancy due to a severe non-CVD related comorbid terminal illness such as cancer;
* No telephone number at which patient can be reached;
* Plans to relocate outside of the NYC area within the next 6 months;
* Inability to communicate over the telephone due to severe cognitive impairment or aphasia.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer P Friedberg, PhD, Principal Investigator — Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY
Locations (1):
- Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a prior American Heart Association-funded study testing the effectiveness of a 6-mo TI vs. AP. Participants were recruited at completion of the AHA study to participate in the current study for an additional 6 months. They continued to receive the intervention to which they were originally assigned in the AHA study.
Groups:
- Tailored Intervention (TI): Tailored phone intervention targeting diet, exercise, and medication adherence based on the transtheoretical model
- Attention Placebo (AP): General phone counseling about health topics unrelated to stroke risk factors (e.g., pain, colorectal cancer screening)
Period: Overall Study
Arm/Group | Tailored Intervention (TI) | Attention Placebo (AP)
Started | 66 | 74
Completed | 63 | 70
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tailored Intervention (TI) | Attention Placebo (AP) | Total
Number analyzed (Participants) | 66 | 74 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.38 (9.86) | 68.73 (10.30) | 67.62 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 64 | 74 | 138
Race/Ethnicity, Customized [Number; unit: participants]
  White (non-Hispanic) | 21 | 27 | 48
  Black/African American (non-Hispanic) | 35 | 34 | 69
  Hispanic/Latino | 6 | 9 | 15
  Other | 3 | 4 | 7
  Refused | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Time Frame: 6 months
Population: restricted to only patients enrolled because they met criteria for high blood pressure at enrollment. Participants were not included if they were did not have elevated blood pressure at enrollment
Measure: Median (Inter-Quartile Range); unit: mm Hg
Arm/Group | Tailored Intervention (TI) | Attention Placebo (AP)
Number analyzed (Participants) | 54 | 59
mm Hg | 130.83 [119.5 to 144.83] | 133.67 [114.5 to 144.0]
Statistical Analysis 1: Comparison: Tailored Intervention (TI) vs Attention Placebo (AP); Robust regressions were performed; Test type: Superiority or Other; p = 0.29, robust regression; controlling for provider clustering

2. Secondary Outcome: Dietary Sodium
Description: self-reported stage of change for adherence to DASH (low-sodium) diet. Pre-action refers to participants reporting that they were in pre-contemplation (no plans to adhere to DASH diet in the next 6 months), contemplation (planning to adhere within the next 6 months) or preparation (planning to adhere within the next month), while action refers to participants reporting that they are in the action stage of change (became adherent to the DASH diet within the past 6 months) and maintenance refers to participants reporting that they are in the maintenance stage of change (became adherent to the DASH diet at least 6 months ago)
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Tailored Intervention (TI) | Attention Placebo (AP)
Number analyzed (Participants) | 63 | 70
participants
  pre-action | 11 | 18
  Action or Maintenance | 52 | 52
Statistical Analysis 1: Comparison: Tailored Intervention (TI) vs Attention Placebo (AP); Test type: Superiority or Other; p = 0.25, Regression, Logistic; This analysis includes participants in pre-action and action/maintenance

3. Secondary Outcome: Total Cholesterol/High Density Lipoprotein Ratio
Time Frame: 6 months
Population: Only participants who provided a blood sample for which cholesterol could be analyzed were included in this analysis
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Tailored Intervention (TI) | Attention Placebo (AP)
Number analyzed (Participants) | 60 | 71
ratio | 3.47 [2.8 to 4.25] | 3.21 [2.8 to 3.81]
Statistical Analysis 1: Comparison: Tailored Intervention (TI) vs Attention Placebo (AP); Test type: Superiority or Other; p = 0.11, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Exercise Adherence
Description: Measured by 7-day Physical Activity Recall
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: hours per week of cardio
Arm/Group | Tailored Intervention (TI) | Attention Placebo (AP)
Number analyzed (Participants) | 63 | 70
hours per week of cardio | 2.50 [1.25 to 5.25] | 2.75 [1 to 6]
Statistical Analysis 1: Comparison: Tailored Intervention (TI) vs Attention Placebo (AP); Test type: Superiority or Other; p = 0.81, Regression, Linear

5. Secondary Outcome: Antihypertensive/ Lipid-lowering Medication Adherence
Description: Measured by Morisky Medication taking questionnaire (self-reported). Scores range from 0-4, with 0 being least adherent and 4 being most adherent
Time Frame: 6 months
Population: One participant in TI did not answer all of the questions on this assessment, so his score could not be computed and therefore he is not included in this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tailored Intervention (TI) | Attention Placebo (AP)
Number analyzed (Participants) | 62 | 70
units on a scale | 3.58 (0.76) | 3.43 (0.79)
Statistical Analysis 1: Comparison: Tailored Intervention (TI) vs Attention Placebo (AP); Test type: Superiority or Other; p = 0.12, Regression, Linear

ADVERSE EVENTS:
Arm/Group | Tailored Intervention (TI) | Attention Placebo (AP)
Serious Adverse Events (participants affected / at risk) | 1/66 | 2/74
Other Adverse Events (participants affected / at risk) | 9/66 | 9/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tailored Intervention (TI) (N=66) | Attention Placebo (AP) (N=74)
Stroke (Nervous system disorders) | 0 | 1
Coronary Artery Bypass Graft (Cardiac disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tailored Intervention (TI) (N=66) | Attention Placebo (AP) (N=74)
Broken bone (Musculoskeletal and connective tissue disorders) | 2 | 2
Torn Ligament (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone/Muscle injury (Musculoskeletal and connective tissue disorders) | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes